CLINICAL TRIAL: NCT03802591
Title: A Multi-Center, Double-Blind, Randomized, Phase III Study of CS1001 in Combination With CAPOX Chemotherapy Compared to Placebo in Combination With CAPOX Chemotherapy in Subjects With Unresectable Locally Advanced or Metastatic GC or GEJ Adenocarcinoma
Brief Title: A Study of CS1001 in Subjects With Gastric Adenocarcinoma or Gastro-Esophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS1001-303
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CS1001 monoclonal antibody (Experimental): in combination with Oxaliplatin and Capecitabine
  Interventions: Drug: CS1001 monoclonal antibody; Drug: Oxaliplatin; Drug: Capecitabine
- CS1001 placebo (Placebo Comparator): in combination with Oxaliplatin and Capecitabine
  Interventions: Drug: CS1001 placebo; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: CS1001 monoclonal antibody — Participant will receive CS1001 monoclonal antibody by intravenous infusion every 3 weeks(Q3W), for up to 24 months
  Arms: CS1001 monoclonal antibody
Drug: CS1001 placebo — Participant will receive CS1001 placebo antibody by intravenous infusion every 3 weeks(Q3W), for up to 24 months
  Arms: CS1001 placebo
Drug: Oxaliplatin — Administered as an IV infusion on Day 1 Q3W
Drug: Capecitabine — Administered by oral, twice a day on Day 1 - Day 14 of each cycle.

SUMMARY:
This is a phase III, multi-Center, randomized, placebo-controlled trial to investigate the efficacy and safety of CS1001 in combination with Oxaliplatin and Capecitabine (CAPOX) chemotherapy in first-line subjects with unresectable locally advanced or metastatic gastric adenocarcinoma (GC) or gastro-esophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years but ≤ 75 years
2. Being able to follow the protocol requirements as per investigator's evaluation.
3. Provide written informed consent before any protocol-related procedure (that is not a part of subject's routine care) is carried out.
4. Unresectable locally advanced or metastatic gastric carcinoma (GC) or gastro-esophageal junction (GEJ) carcinoma, and have histologically confirmed predominant adenocarcinoma.
5. The subject may have at least a measurable lesion or an evaluable lesion, if not measurable; the investigator will carry out evaluation according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 within 28 days prior to randomization.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
7. Expected survival ≥ 3 months.
8. Subject must not have received systemic treatment (including HER2 inhibitor) for advanced or metastatic gastric carcinoma.
9. Subject must provide tumor tissue samples for biomarker analysis in order to determine the expression of PD-L1. According to central laboratory test, the PD-L1 expression is ≥ 5% in tumor tissue (including PD-L1 expression in tumor cells and tumor infiltrating immune cells).
10. Permitted prior treatment: Subjects with GC or GEJ carcinoma priorly treated with adjuvant or neoadjuvant therapy, who experience clinical progression of disease at least 6 months after last dose are allowed to be enrolled.
11. Subjects must have adequate organ function as assessed in the laboratory tests
12. Subjects with active hepatitis B or active hepatitis C must receive antiviral treatment for at least 14 days prior to the first dose of study treatment and pass the hepatitis B virus (HBV) DNA titer test (≤ 500 IU/mL or 2500 copies/mL) and hepatitis C virus (HCV) RNA test (≤ lower limit of detection) before being enrolled. The subject should be willing to continue effective anti-viral treatment during the study.
13. Female subject with childbearing potential must have negative serum pregnancy test result at screening, except for those with available sterilization operation record or post-menopausal subjects. Female subject with childbearing potential or male subjects and their partners must agree to take effective contraceptive measures from the day of signing ICF till at least 6 months after the last dosing of investigational product.

Exclusion Criteria:

1. Known HER-2 positivity.
2. A known additional primary malignancy that occurred within 5 years prior to the first dose of investigational treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
3. Known primary central nerve system (CNS) tumor or meningeal metastasis, or unstable CNS metastasis (symptomatic within 4 weeks before first dose of investigational product, requiring corticosteroid treatment, or without radiologic evidence supporting stable status for over 4 weeks prior to the first dose of investigational product).
4. Any severe or uncontrolled systemic disease, for example diabetes mellitus or hypertension, that may increase the risk associated with participation or investigational product administration, or compromise subject's ability to receive investigational product, as per investigator's judgment.
5. Known positive human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS).
6. Has had prior chemotherapy, immune therapy, biological therapy (including cancer vaccine, cytokine therapy or growth factors to control cancer) used as systemic treatment for cancer, within 14 days before the first dose of investigational product.
7. Any prior treatment of antibody/drug that targets at T-cell coregulatory proteins or immune checkpoints pathways(including anti-PD-1, anti-PD-L1, anti-CTLA4, anti-TIM3, anti-LAG3 antibody, etc.).
8. Subjects with conditions that in the investigator's opinion are not suitable for participating in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) evaluated by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | from the date of randomization to the first date of recorded progression or all-cause death, whichever comes first, assessed up to approximately 27 months
Overall survival (OS) | from the date of randomization to the first date of recorded all-cause death, assessed up to approximately 38 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) evaluated by Blinded Independent Central Review Committee (BICR) according to RECIST v1.1 | from the date of randomization to the first date of recorded progression or all-cause death, whichever comes first, assessed up to approximately 27 months
Objective response rate (ORR) evaluated by investigators according to RECIST v1.1 | from the first dose of treatment until the best response, assessed up to 27 months
Duration of response (DOR) (evaluated by investigators according to RECIST v1.1) | from date of first documented objective response until first documented sign of disease progression or death due to any causes, whichever comes first, assessed up to approximately 27 months
Overall survival rate at 12 months and 24 months | from the date of randomization to the first date of recorded all-cause death, assessed up to approximately 38 months
Evaluate the safety of CS1001 in combination with CAPOX chemotherapy compared to placebo in combination with CAPOX chemotherapy | from the date of randomization to the first date of recorded all-cause death, assessed up to approximately 38 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

REFERENCES:
- [Derived] Zhang X, Wang J, Wang G, Zhang Y, Fan Q, Lu C, Hu C, Sun M, Wan Y, Sun S, Wang J, Zhang L, Shu Y, Luo J, Zhu D, Shen Z, Yao S, Shi Q, Yang J, Shen L; GEMSTONE-303 Investigators. First-Line Sugemalimab Plus Chemotherapy for Advanced Gastric Cancer: The GEMSTONE-303 Randomized Clinical Trial. JAMA. 2025 Apr 15;333(15):1305-1314. doi: 10.1001/jama.2024.28463. PMID 39992668